CLINICAL TRIAL: NCT06878833
Title: A Multidose, Randomized, Double-Blind Study to Evaluate the Safety and Tolerability of Long-Acting Oral Risperidone (LYN-005) in Participants With Schizophrenia or Schizoaffective Disorder
Brief Title: A Study to Evaluate the Safety and Tolerability of Long-Acting Oral Risperidone (LYN-005) in Participants With Schizophrenia or Schizoaffective Disorder
Acronym: Starlyng-2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor stopped operations
Sponsor: Lyndra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LYN-005-C-302
Record Dates: First submitted 2025-02-25; First posted 2025-03-17 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Risperidone; LYN-005; long-acting oral (LAO) therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open Label (OL) Cohort (Experimental): After a 7-day run-in period in which participants receive immediate release (IR) risperidone (2 mg/day, 4 mg/day, or 6 mg/day, based on prior antipsychotic drug dose) and a single dose of LYN-005-matched placebo, participants receive weekly doses of 15, 30, or 45 mg of LYN-005 for 7 weeks.
  Interventions: Drug: LYN-005 (risperidone); Drug: Placebo for LYN-005; Drug: IR Risperidone
- Double Blind (DB) Cohort: LYN-005 (Experimental): After a 7-day run-in period in which participants receive IR risperidone (2 mg/day, 4 mg/day, or 6 mg/day, based on prior antipsychotic drug dose) and a single dose of LYN-005-matched placebo, participants receive weekly doses of 15, 30, or 45 mg of LYN-005 and daily doses of IR risperidone-matched placebo for 26 weeks.
  Interventions: Drug: LYN-005 (risperidone); Drug: Placebo for LYN-005; Drug: IR Risperidone; Drug: Placebo for IR Risperidone
- Double Blind (DB) Cohort: IR Risperidone (Active Comparator): After a 7-day run-in period in which participants receive IR risperidone (2 mg/day, 4 mg/day, or 6 mg/day, based on prior antipsychotic drug dose) and a single dose of LYN-005-matched placebo, participants receive daily doses of 2, 4, or 6 mg IR risperidone and weekly doses of LYN-005-matched placebo for 26 weeks.
  Interventions: Drug: Placebo for LYN-005; Drug: IR Risperidone; Drug: Placebo for IR Risperidone

INTERVENTIONS:
Drug: LYN-005 (risperidone) — long-acting oral (LAO) capsule
  Arms: Double Blind (DB) Cohort: LYN-005; Open Label (OL) Cohort
Drug: Placebo for LYN-005 — capsule
Drug: IR Risperidone — tablets
Drug: Placebo for IR Risperidone — tablets
  Arms: Double Blind (DB) Cohort: IR Risperidone; Double Blind (DB) Cohort: LYN-005

SUMMARY:
Lyndra Therapeutics, Inc., is developing a long-acting oral (LAO) treatment of risperidone (LYN-005) in a capsule dosage form (LYNX® drug delivery platform). The intent of LYN-005 is to reduce the dosing frequency of orally-administered risperidone to once weekly or less and, thereby improve treatment adherence and management of schizophrenia and schizoaffective disorder.

This study will evaluate the safety and tolerability of multiple administrations of LYN-005 at 3 dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 and ≤65 years.
2. Current diagnosis of schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria as confirmed by the Mini International Neuropsychiatric Interview version 7.0.2 (MINI 7.0.2).
3. Psychiatric criteria:

   1. Duration of diagnosis of schizophrenia or schizoaffective disorder for ≥2 years.
   2. Outpatient; not hospitalized for worsening of schizophrenia within the last 6 months (partial hospitalization for social management within this time period is acceptable).
   3. Medically stable over the last month and psychiatrically stable without significant symptom exacerbation over the last 3 months.
4. Stabilized on a therapeutic dose of an oral antipsychotic drug for a minimum of 6 weeks at the time of Screening.
5. On a stable dosage of all permitted non-antipsychotic medications (except for medication to be used on an as-needed basis) for at least 1 month before the Screening visit and for the duration of the study.
6. Clinical Global Impression-Severity (CGI-S) score of ≤4 (moderately ill) at Screening and Day -7.
7. Positive and Negative Syndrome Scale (PANSS) score of ≤80 points at Screening.
8. Body mass index (BMI) of ≥18 kg/m2 and ≤38 kg/m2.
9. Able to read and understand study procedures and provide written informed consent before the initiation of any protocol-specific procedures.
10. Willing to comply with all protocol-specified procedures and availability for the duration of the study.

Exclusion Criteria:

1. Participants with known clinically significant esophageal or GI disease, including but not limited to:

   1. Known strictures such as esophageal web, pyloric stenosis, or small intestinal stricture, or participants with high risk of stricture, e.g., Crohn's disease.
   2. Prior varices or small or large bowel obstructions.
   3. Prior abdominal or upper gastrointestinal surgery including gastric bypass or removal of a significant portion of the gastrointestinal (GI) tract that may impose a high risk of strictures (prior uncomplicated laparoscopic procedures including appendectomy or colectomy are permitted).
   4. History of diarrhea or constipation within 3 months of Screening that in the opinion of the investigator would be considered clinically significant.
   5. Multiple episodes of moderate or severe abdominal pain within 3 months of Screening.
   6. History of moderate to severe Acid Reflux Disease or a score of ≥2 on the Acid Reflux Severity Scale (ARSS) [2], indicating moderate to severe symptoms.
2. PILL-5 questionnaire score of 5 or greater.
3. Any clinically significant medical, surgical or psychiatric condition that in the opinion of the investigator would exclude them from the study, including:

   1. Presence of an uncontrolled, unstable, clinically significant medical condition that could put the participant at risk because of participation in the study, interfere with the participant's ability to participate in the study or influence the interpretation of safety or pharmacokinetic (PK) evaluations.
   2. History of a major cardiovascular event (myocardial infarction, cardiac surgery or revascularization, unstable angina, stroke, or transient ischemic attack) or a hospitalization for heart failure within 6 months of Screening.
   3. Any clinically significant illness, medical or surgical procedure or trauma within 4 weeks of Screening.
   4. Known immunocompromised status, including individuals who have undergone organ transplantation, on immunosuppression for an immune mediated disease, or are positive for human immunodeficiency virus (HIV).
   5. Positive test for active hepatitis B or C at Screening. Participants with successfully treated hepatitis B infection which has been resolved for greater than 1 year or successfully treated hepatitis C infection will not be excluded.
   6. Have donated more than 250 mL of blood within 30 days of Screening.
   7. Have difficulties with venipuncture/cannulation, including difficulty accessing veins for blood sampling and/or history of coagulopathy or endocarditis.
   8. Current DSM-5 diagnosis of major depressive episode, panic disorder, agoraphobia, social anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder on the MINI 7.0.2 or in the judgment of the Investigator. (Note that individuals with depression secondary to schizoaffective disorder are eligible).
   9. Suicidal ideation associated with actual intent and a method or plan in the past 6 months, as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS; i.e., "Yes" answers on items 4 or 5) at Screening and Day -7or having made a suicide attempt within the last 2 years.
   10. Known or suspected (non-febrile) seizure disorder.
   11. History of neuroleptic malignant syndrome
   12. Current or history of clinically significant tardive dyskinesia.
   13. Known or suspected diagnosis of intellectual disability or organic brain disorder or other diagnosis that is primarily responsible for current symptoms and functional impairment.
   14. Medically non-adherent in the management of their schizophrenia/schizoaffective disorder.
4. Use of the below medications/treatments in the 2 weeks before enrollment:

   1. Proton pump inhibitors or H2 blockers.
   2. Prokinetic agents.
   3. Medications that may interfere with the absorption, metabolism, or excretion of risperidone, e.g.: i. Drugs metabolized via Cytochrome P450 3A4 (CYP3A4) pathway, such as macrolide antibiotics and azole antifungals; ii. Moderate or strong CYP3A4 p-glycoprotein (P-gp) enzyme inducers and inhibitors (carbamazepine, phenytoin, rifampicin, phenobarbital, itraconazole, verapamil); iii. Moderate or strong Cytochrome P450 2D6 (CYP2D6) inhibitors (e.g., fluoxetine, fluoxetine combinations, paroxetine, or quinidine).
   4. Concomitant medications, natural remedies, supplements, or vitamins that are associated with changes to gastric motility or pH. Use of antacids is permissible, except within 2 hours of dosing with LYN-005.
   5. Use of more than one antidepressant for the treatment of depression; or if on just one, a change in dose within 6 weeks of Screening.
   6. Depot antipsychotic use within 6 months of Screening.
   7. Electroconvulsive therapy within 3 months of Screening.
5. Participants with clinically significant abnormal safety (e.g. physical examination, vital sign) or safety laboratory assessments, specifically:

   1. Presence of a clinically significant abnormal laboratory result on blood or urine safety tests at Screening.
   2. Anemia (hemoglobin below lower limit of normal reference range) at Screening.
   3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≥3.0 × upper limit of normal (ULN), or total bilirubin ≥1.5 × ULN.
   4. Moderate or severe renal insufficiency at Screening (glomerular filtration rate <60 mL/min, as determined the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation).
   5. Heart rate of <50 beats per minute (bpm) at Screening.
   6. Systolic blood pressure <100 or ≥150 mmHg and/or diastolic blood pressure <60 mmHg or ≥100 mmHg, and/or orthostatic hypotension, at Screening.
   7. HbA1c ≥6.5% at Screening.
   8. Positive fecal occult blood test at Screening.
   9. Clinically significant prolactin elevation (≥200 ng/mL for females; ≥100 ng/mL for males).
6. The following specified patterns of substance use at Screening:

   1. Fulfillment of the DSM-5 criteria for moderate or severe substance use disorder (excluding nicotine and caffeine) within 6 months of Screening.
   2. History of alcohol consumption exceeding moderate use; in males exceeding 21 units per week and in females exceeding 14 units per week (1 unit = 360 ml beer, 25 mL of 40% spirit or a 125 mL glass of wine) over the past month. Participants are not permitted to consume alcohol during the inpatient stay nor 12 hours before any clinic visit while outpatient.
   3. Positive ethanol breathalyzer.
   4. Positive urine drug screen for substances of abuse other than cannabis at screening or Day -7.
   5. Heavy nicotine use (consumption of >40 cigarettes or >36 mg of nicotine from other sources [e.g., vaping products] daily) or daily use of smokeless tobacco.
7. Participants of reproductive potential who are (hetero) sexually active but unwilling to use acceptable means of contraception through the End-of-Study. For clarity, participants who are at least 1 year post-menopausal are not of reproductive potential. Acceptable means of contraception include:

   1. Participants who have been surgically sterilized.
   2. Females of reproductive potential: diaphragm, injectable, oral/patch contraceptives for a minimum of 6 weeks, contraceptive sponge, implant, or intrauterine device in use prior to enrollment.
   3. Males: condom in combination with any of the above means of contraception.
   4. All participants: abstinence may be an acceptable means of contraception as long as the individual consents to initiate immediate use of double barrier protection for the duration of the study should (hetero) sexual intercourse occur.
8. Participants who are nursing or who have positive or indeterminate pregnancy tests at either Screening (serum test) or Day -7 (urine test).
9. Participants with history of X-ray, computed tomography (CT) scan or angiogram of the abdomen within one year of Screening
10. Use of any experimental agent within 1 month or 5 half-lives of Screening, whichever is longer.
11. Employee or immediate family member of employees of the site, Sponsor, or study-related vendors.
12. History of a serious allergic or hypersensitivity reaction to risperidone or LYN-005 excipients (refer to Investigator's Brochure). Previous use of LYN-005 alone, does not exclude participants.
13. CYP2D6 poor or indeterminate metabolizer status based on genetic testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-18 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | OL Cohort: Screening through Day 57; DB Cohort: Screening through Day 203

SECONDARY OUTCOMES:
PK Evaluation: Minimum Observed Concentration (Cmin) of Active Moiety at Week 5 (OL Cohort only) | Week 5: postdose: 24 hours (±30 minutes), 48 hours (±30 minutes), 72 hours (±30 minutes), 96 hours (±30 minutes), 120 hours (±30 minutes),144 hours (±30 minutes), and 168 hours (up to 30 minutes before 168 hours)
PK Evaluation: Maximal Observed Concentration (Cmax) of Active Moiety at Week 5 (OL Cohort only) | Week 5: postdose: 24 hours (±30 minutes), 48 hours (±30 minutes), 72 hours (±30 minutes), 96 hours (±30 minutes), 120 hours (±30 minutes),144 hours (±30 minutes), and 168 hours (up to 30 minutes before 168 hours)
PK Evaluation: Average Concentration (Cavg) of Active Moiety at Week 5 (OL Cohort only) | Week 5: postdose: 24 hours (±30 minutes), 48 hours (±30 minutes), 72 hours (±30 minutes), 96 hours (±30 minutes), 120 hours (±30 minutes),144 hours (±30 minutes), and 168 hours (up to 30 minutes before 168 hours)
Change in Structured Clinical Interview for the Positive and Negative Syndrome Scale (SCI-PANSS) Over Time | OL Cohort: Baseline, Day 22 and 43; DB Cohort: Baseline, Days 22, 43, 92, 106, 134, 162, 183

CONTACTS AND LOCATIONS:
Overall Officials: Nayana Nagaraj, Study Director — Lyndra Inc.

IPD SHARING:
Plan to Share IPD: No